CLINICAL TRIAL: NCT00318331
Title: Randomized Clinical Trial Comparing Enteral Glutamine Supplementation to Standard of Care Enteral Feeding in Critical Illness
Brief Title: Enteral Glutamine in Critical Illness
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to meet enrollment numbers
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Dr. Michael DePietro, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Glutamine
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Critical Illness; Sepsis; Respiratory Insufficiency
Keywords: Glutamine; Critical Illness; Enteral Feeding; Blood Volume Analysis
MeSH Terms: conditions — Critical Illness; Sepsis; Respiratory Insufficiency | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Will receive enteral glutamine
  Interventions: Drug: Glutamine
- B (No Intervention): No enteral glutamine given

INTERVENTIONS:
Drug: Glutamine — Group A patients will receive 0.5g/kg/day of enteral glutamine daily while they are receiving tube feeds or at the end of 28 days (whichever comes first)
  Arms: A

SUMMARY:
Glutamine is an amino acid which is rapidly depleted in critical illness. It is used as energy by cells that line the gut, vital for immune system function, and works as an anti-oxidant. Glutamine supplementation has been shown to improve outcomes in ICU patients. We hypothesize that critically ill patients given extra glutamine will have less of an inflammatory response and therefore better outcomes than patients not given extra glutamine. Our study randomizes patients to tube feeding with OR without extra glutamine to see if it affects patient outcomes as well as markers of inflammation.

DETAILED DESCRIPTION:
Glutamine, a nonessential amino acid, is preferred fuel for rapidly proliferating cells in human body. Those cells include the enterocytes in small intestine, lymphocytes, macrophages, and fibroblasts. Glutamine also transports nitrogen between tissues and serves as a precursor to glutathione which is a potent antioxidant. A healthy human body contains abundant glutamine, either from diet or from skeletal muscle tissue that synthesizes it.

During critical illness the demand for glutamine is increased. Rapid depletion of glutamine stores in critically ill patients has been described and correlated to increased mortality. Glutamine depletion may be deleterious in critical illness because of adverse effects on the essential functions mentioned above. For example glutamine depletion may cause gut mucosal barrier function to deteriorate, leading to bacterial translocation and enhanced systemic inflammatory response with increased risk for multisystem organ failure. Clinical trials performed in a wide range of patients with serious illness, including cancer, trauma, burn, major surgery and critical illness, have demonstrated possible benefits of glutamine supplementation. Interpretation of the results of multiple studies is made difficult based on differences in glutamine dosing, route of administration, population studied, and endpoints used.

Blood volume analysis has been shown to be a good measure of capillary leak. The DAXOR blood volume analyzer kit was recently approved by the FDA for blood volume analyses and also has the capacity of measuring capillary permeability by looking at the slope of albumin transudation. It is a simpler way to measure capillary permeability than other methods described.

Reviewing the previous study results, glutamine supplementation in parental form and with higher dose in various patient populations has shown evidence of being beneficial. Studies of enteral glutamine therapy have also showed benefits, but results are less consistent possibly because of the heterogeneous study methodology described above. Moreover, most of the studies are carried out in burn patients and surgical patients; there were few studies in critical ill medical patients. Finally no study has specifically looked at the mechanism via which glutamine has conferred protection.

Comparison: Critically ill patients given enteral tube feeds compared to critically ill patients given enteral tube feeds with supplemental glutamine.

ELIGIBILITY:
Inclusion Criteria:

* Admission to MICU/ CICU
* Age greater than or equal to 18 years old
* Requirement for enteral nutrition
* Presence or planned insertion of central venous catheter as part of routine medical care
* Requirement for mechanical ventilation
* APACHE II Score >/= 15

Exclusion Criteria:

* Female of child-bearing age (i.e. less than 45 years old)
* Enteral nutrition begun prior to randomization
* Receiving Total Parenteral Nutrition
* Requirement for protein restriction
* Creatinine >4 mg/dl
* History of cirrhosis and/or clinical signs of heptic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
Length of ICU stay | 28 days
Number of Ventilator Days | 28 days
Number of days receiving antibiotics | 28 days

SECONDARY OUTCOMES:
Change in APACHE Score | 72 hours
Change in Number of SIRS Criteria | 72 hours
Change in Capillary Leak as measured by blood volume analysis | 72 hours
Change in CRP | 72 hours
Correlation between capillary permeability and APACHE Score | 72 hours
Correlation between capillary permeability and Mortality | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael DePietro, M.D., Principal Investigator
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

REFERENCES:
- [Background] Souba WW, Smith RJ, Wilmore DW. Glutamine metabolism by the intestinal tract. JPEN J Parenter Enteral Nutr. 1985 Sep-Oct;9(5):608-17. doi: 10.1177/0148607185009005608. No abstract available. PMID 3900455
- [Background] Gamrin L, Essen P, Forsberg AM, Hultman E, Wernerman J. A descriptive study of skeletal muscle metabolism in critically ill patients: free amino acids, energy-rich phosphates, protein, nucleic acids, fat, water, and electrolytes. Crit Care Med. 1996 Apr;24(4):575-83. doi: 10.1097/00003246-199604000-00005. PMID 8612406
- [Background] Conejero R, Bonet A, Grau T, Esteban A, Mesejo A, Montejo JC, Lopez J, Acosta JA. Effect of a glutamine-enriched enteral diet on intestinal permeability and infectious morbidity at 28 days in critically ill patients with systemic inflammatory response syndrome: a randomized, single-blind, prospective, multicenter study. Nutrition. 2002 Sep;18(9):716-21. doi: 10.1016/s0899-9007(02)00847-x. PMID 12297203
- [Background] Oudemans-van Straaten HM, Bosman RJ, Treskes M, van der Spoel HJ, Zandstra DF. Plasma glutamine depletion and patient outcome in acute ICU admissions. Intensive Care Med. 2001 Jan;27(1):84-90. doi: 10.1007/s001340000703. PMID 11280678
- [Background] Planas M, Schwartz S, Arbos MA, Farriol M. Plasma glutamine levels in septic patients. JPEN J Parenter Enteral Nutr. 1993 May-Jun;17(3):299-300. doi: 10.1177/0148607193017003299. No abstract available. PMID 8505843
- [Background] Ziegler TR, Young LS, Benfell K, Scheltinga M, Hortos K, Bye R, Morrow FD, Jacobs DO, Smith RJ, Antin JH, et al. Clinical and metabolic efficacy of glutamine-supplemented parenteral nutrition after bone marrow transplantation. A randomized, double-blind, controlled study. Ann Intern Med. 1992 May 15;116(10):821-8. doi: 10.7326/0003-4819-116-10-821. PMID 1567096
- [Background] Griffiths RD, Jones C, Palmer TE. Six-month outcome of critically ill patients given glutamine-supplemented parenteral nutrition. Nutrition. 1997 Apr;13(4):295-302. PMID 9178278
- [Background] Wischmeyer PE, Lynch J, Liedel J, Wolfson R, Riehm J, Gottlieb L, Kahana M. Glutamine administration reduces Gram-negative bacteremia in severely burned patients: a prospective, randomized, double-blind trial versus isonitrogenous control. Crit Care Med. 2001 Nov;29(11):2075-80. doi: 10.1097/00003246-200111000-00006. PMID 11700398
- [Background] Wischmeyer PE. Clinical applications of L-glutamine: past, present, and future. Nutr Clin Pract. 2003 Oct;18(5):377-85. doi: 10.1177/0115426503018005377. PMID 16215069
- [Background] Garrel D, Patenaude J, Nedelec B, Samson L, Dorais J, Champoux J, D'Elia M, Bernier J. Decreased mortality and infectious morbidity in adult burn patients given enteral glutamine supplements: a prospective, controlled, randomized clinical trial. Crit Care Med. 2003 Oct;31(10):2444-9. doi: 10.1097/01.CCM.0000084848.63691.1E. PMID 14530749
- [Background] Oberhoffer M, Karzai W, Meier-Hellmann A, Bogel D, Fassbinder J, Reinhart K. Sensitivity and specificity of various markers of inflammation for the prediction of tumor necrosis factor-alpha and interleukin-6 in patients with sepsis. Crit Care Med. 1999 Sep;27(9):1814-8. doi: 10.1097/00003246-199909000-00018. PMID 10507603
- [Background] Lobo SM, Lobo FR, Bota DP, Lopes-Ferreira F, Soliman HM, Melot C, Vincent JL. C-reactive protein levels correlate with mortality and organ failure in critically ill patients. Chest. 2003 Jun;123(6):2043-9. doi: 10.1378/chest.123.6.2043. PMID 12796187
- [Background] Singleton KD, Serkova N, Beckey VE, Wischmeyer PE. Glutamine attenuates lung injury and improves survival after sepsis: role of enhanced heat shock protein expression. Crit Care Med. 2005 Jun;33(6):1206-13. doi: 10.1097/01.ccm.0000166357.10996.8a. PMID 15942332
- [Background] Wischmeyer PE. Can glutamine turn off the motor that drives systemic inflammation? Crit Care Med. 2005 May;33(5):1175-8. doi: 10.1097/01.ccm.0000162686.28604.81. No abstract available. PMID 15891373
- [Background] De-Souza DA, Greene LJ. Intestinal permeability and systemic infections in critically ill patients: effect of glutamine. Crit Care Med. 2005 May;33(5):1125-35. doi: 10.1097/01.ccm.0000162680.52397.97. PMID 15891348
- [Background] Preiser JC, Coeffier M. Heme oxygenase: a new piece in the glutamine puzzle. Crit Care Med. 2005 Feb;33(2):457-8. doi: 10.1097/01.ccm.0000153412.49304.22. No abstract available. PMID 15699860
- [Background] Choudhry MA, Haque F, Khan M, Fazal N, Al-Ghoul W, Ravindranath T, Gamelli RL, Sayeed MM. Enteral nutritional supplementation prevents mesenteric lymph node T-cell suppression in burn injury. Crit Care Med. 2003 Jun;31(6):1764-70. doi: 10.1097/01.CCM.0000063053.31485.DF. PMID 12794418
- [Background] Goeters C, Wenn A, Mertes N, Wempe C, Van Aken H, Stehle P, Bone HG. Parenteral L-alanyl-L-glutamine improves 6-month outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2032-7. doi: 10.1097/00003246-200209000-00013. PMID 12352037
- [Background] Novak F, Heyland DK, Avenell A, Drover JW, Su X. Glutamine supplementation in serious illness: a systematic review of the evidence. Crit Care Med. 2002 Sep;30(9):2022-9. doi: 10.1097/00003246-200209000-00011. PMID 12352035
- [Background] Berard MP, Zazzo JF, Condat P, Vasson MP, Cynober L. Total parenteral nutrition enriched with arginine and glutamate generates glutamine and limits protein catabolism in surgical patients hospitalized in intensive care units. Crit Care Med. 2000 Nov;28(11):3637-44. doi: 10.1097/00003246-200011000-00016. PMID 11098966
- [Background] Beale RJ, Bryg DJ, Bihari DJ. Immunonutrition in the critically ill: a systematic review of clinical outcome. Crit Care Med. 1999 Dec;27(12):2799-805. doi: 10.1097/00003246-199912000-00032. PMID 10628629
- [Background] Coeffier M, Dechelotte P. The role of glutamine in intensive care unit patients: mechanisms of action and clinical outcome. Nutr Rev. 2005 Feb;63(2):65-9. doi: 10.1111/j.1753-4887.2005.tb00123.x. PMID 15762090
- [Background] Heyland DK, Dhaliwal R, Drover JW, Gramlich L, Dodek P; Canadian Critical Care Clinical Practice Guidelines Committee. Canadian clinical practice guidelines for nutrition support in mechanically ventilated, critically ill adult patients. JPEN J Parenter Enteral Nutr. 2003 Sep-Oct;27(5):355-73. doi: 10.1177/0148607103027005355. PMID 12971736
- [Background] Wischmeyer PE, Riehm J, Singleton KD, Ren H, Musch MW, Kahana M, Chang EB. Glutamine attenuates tumor necrosis factor-alpha release and enhances heat shock protein 72 in human peripheral blood mononuclear cells. Nutrition. 2003 Jan;19(1):1-6. doi: 10.1016/s0899-9007(02)00839-0. PMID 12507630
- [Background] Chwals WJ. Regulation of the cellular and physiological effects of glutamine. Mini Rev Med Chem. 2004 Oct;4(8):833-8. doi: 10.2174/1389557043403396. PMID 15544544
- [Background] Bistrian BR. Practical recommendations for immune-enhancing diets. J Nutr. 2004 Oct;134(10 Suppl):2868S-2872S; discussion 2895S. doi: 10.1093/jn/134.10.2868S. PMID 15465803
- [Background] Baudouin SV, Evans TW. Nutritional support in critical care. Clin Chest Med. 2003 Dec;24(4):633-44. doi: 10.1016/s0272-5231(03)00101-1. PMID 14710695
- [Background] Hall JC, Dobb G, Hall J, de Sousa R, Brennan L, McCauley R. A prospective randomized trial of enteral glutamine in critical illness. Intensive Care Med. 2003 Oct;29(10):1710-6. doi: 10.1007/s00134-003-1937-2. Epub 2003 Aug 16. PMID 12923621
- [Background] Garcia-de-Lorenzo A, Zarazaga A, Garcia-Luna PP, Gonzalez-Huix F, Lopez-Martinez J, Mijan A, Quecedo L, Casimiro C, Usan L, del Llano J. Clinical evidence for enteral nutritional support with glutamine: a systematic review. Nutrition. 2003 Sep;19(9):805-11. doi: 10.1016/s0899-9007(03)00103-5. PMID 12921894
- [Background] Sacks GS, Genton L, Kudsk KA. Controversy of immunonutrition for surgical critical-illness patients. Curr Opin Crit Care. 2003 Aug;9(4):300-5. doi: 10.1097/00075198-200308000-00008. PMID 12883285
- [Background] Wernerman J. Glutamine and acute illness. Curr Opin Crit Care. 2003 Aug;9(4):279-85. doi: 10.1097/00075198-200308000-00005. PMID 12883282
- [Background] Oehler R, Roth E. Regulative capacity of glutamine. Curr Opin Clin Nutr Metab Care. 2003 May;6(3):277-82. doi: 10.1097/01.mco.0000068962.34812.ac. PMID 12690259
- [Background] Kelly D, Wischmeyer PE. Role of L-glutamine in critical illness: new insights. Curr Opin Clin Nutr Metab Care. 2003 Mar;6(2):217-22. doi: 10.1097/00075197-200303000-00011. PMID 12589192
- [Background] Koretz RL. Immunonutrition: fact, fantasy, and future. Curr Gastroenterol Rep. 2002 Aug;4(4):332-7. doi: 10.1007/s11894-002-0084-1. PMID 12149179
- [Background] Andrews F, Griffiths R. Glutamine-enhanced nutrition in the critically ill patient. Hosp Med. 2002 Mar;63(3):144-7. doi: 10.12968/hosp.2002.63.3.2058. PMID 11933816
- [Background] Oehler R, Pusch E, Dungel P, Zellner M, Eliasen MM, Brabec M, Roth E. Glutamine depletion impairs cellular stress response in human leucocytes. Br J Nutr. 2002 Jan;87 Suppl 1:S17-21. doi: 10.1079/bjn2001453. PMID 11895151
- [Background] Andrews FJ, Griffiths RD. Glutamine: essential for immune nutrition in the critically ill. Br J Nutr. 2002 Jan;87 Suppl 1:S3-8. doi: 10.1079/bjn2001451. PMID 11895153
- [Background] Velasco N, Hernandez G, Wainstein C, Castillo L, Maiz A, Lopez F, Guzman S, Bugedo G, Acosta AM, Bruhn A. Influence of polymeric enteral nutrition supplemented with different doses of glutamine on gut permeability in critically ill patients. Nutrition. 2001 Nov-Dec;17(11-12):907-11. doi: 10.1016/s0899-9007(01)00613-x. PMID 11744338
- [Background] Griffiths RD. The evidence for glutamine use in the critically-ill. Proc Nutr Soc. 2001 Aug;60(3):403-10. doi: 10.1079/pns200197. PMID 11681816
- [Background] Heyland DK, Novak F, Drover JW, Jain M, Su X, Suchner U. Should immunonutrition become routine in critically ill patients? A systematic review of the evidence. JAMA. 2001 Aug 22-29;286(8):944-53. doi: 10.1001/jama.286.8.944. PMID 11509059
- [Background] Labow BI, Souba WW. Glutamine. World J Surg. 2000 Dec;24(12):1503-13. doi: 10.1007/s002680010269. PMID 11193715
- [Background] Barbosa E, Moreira EA, Goes JE, Faintuch J. Pilot study with a glutamine-supplemented enteral formula in critically ill infants. Rev Hosp Clin Fac Med Sao Paulo. 1999 Jan-Feb;54(1):21-4. doi: 10.1590/s0041-87811999000100005. PMID 10488597
- [Background] Mittendorfer B, Gore DC, Herndon DN, Wolfe RR. Accelerated glutamine synthesis in critically ill patients cannot maintain normal intramuscular free glutamine concentration. JPEN J Parenter Enteral Nutr. 1999 Sep-Oct;23(5):243-50; discussion 250-2. doi: 10.1177/0148607199023005243. PMID 10485436
- [Background] Saito H, Furukawa S, Matsuda T. Glutamine as an immunoenhancing nutrient. JPEN J Parenter Enteral Nutr. 1999 Sep-Oct;23(5 Suppl):S59-61. doi: 10.1177/014860719902300515. PMID 10483897
- [Background] Sacks GS. Glutamine supplementation in catabolic patients. Ann Pharmacother. 1999 Mar;33(3):348-54. doi: 10.1345/aph.18200. PMID 10200861
- [Background] Jones C, Palmer TE, Griffiths RD. Randomized clinical outcome study of critically ill patients given glutamine-supplemented enteral nutrition. Nutrition. 1999 Feb;15(2):108-15. doi: 10.1016/s0899-9007(98)00172-5. PMID 9990574
- [Background] Jackson NC, Carroll PV, Russell-Jones DL, Sonksen PH, Treacher DF, Umpleby AM. The metabolic consequences of critical illness: acute effects on glutamine and protein metabolism. Am J Physiol. 1999 Jan;276(1):E163-70. doi: 10.1152/ajpendo.1999.276.1.E163. PMID 9886963
- [Background] Griffiths RD. Outcome of critically ill patients after supplementation with glutamine. Nutrition. 1997 Jul-Aug;13(7-8):752-4. doi: 10.1016/s0899-9007(97)83039-0. PMID 9263282
- [Background] van der Hulst RR, von Meyenfeldt MF, Soeters PB. Glutamine: an essential amino acid for the gut. Nutrition. 1996 Nov-Dec;12(11-12 Suppl):S78-81. doi: 10.1016/s0899-9007(97)85206-9. PMID 8974125
- [Background] Heberer M, Babst R, Juretic A, Gross T, Horig H, Harder F, Spagnoli GC. Role of glutamine in the immune response in critical illness. Nutrition. 1996 Nov-Dec;12(11-12 Suppl):S71-2. doi: 10.1016/s0899-9007(97)85203-3. PMID 8974122
- [Background] Jensen GL, Miller RH, Talabiska DG, Fish J, Gianferante L. A double-blind, prospective, randomized study of glutamine-enriched compared with standard peptide-based feeding in critically ill patients. Am J Clin Nutr. 1996 Oct;64(4):615-21. doi: 10.1093/ajcn/64.4.615. PMID 8839508
- [Background] MacFie J, O'Boyle C, Mitchell CJ, Buckley PM, Johnstone D, Sudworth P. Gut origin of sepsis: a prospective study investigating associations between bacterial translocation, gastric microflora, and septic morbidity. Gut. 1999 Aug;45(2):223-8. doi: 10.1136/gut.45.2.223. PMID 10403734
- [Background] Preiser JC, Wernerman J. Glutamine, a life-saving nutrient, but why? Crit Care Med. 2003 Oct;31(10):2555-6. doi: 10.1097/01.CCM.0000084863.47943.6F. No abstract available. PMID 14530768
- [Background] Rector WG Jr, Ibarra F. Intravascular volume in cirrhosis. Reassessment using improved methodology. Dig Dis Sci. 1988 Apr;33(4):460-6. doi: 10.1007/BF01536032. PMID 3349893
- [Background] Haraldsson B, Rippe B. Influence of perfusate oncotic pressure on the transcapillary clearance of albumin in maximally vasodilated rat skeletal muscle. Acta Physiol Scand. 1987 Jun;130(2):219-28. doi: 10.1111/j.1748-1716.1987.tb08131.x. PMID 3604712
- [Background] Margarson MP, Soni NC. Effects of albumin supplementation on microvascular permeability in septic patients. J Appl Physiol (1985). 2002 May;92(5):2139-45. doi: 10.1152/japplphysiol.00201.2001. PMID 11960967
- [Background] Alrawi SJ, Miranda LS, Cunningham JN Jr, Acinapura AJ, Raju R. Correlation of blood volume values and pulmonary artery catheter measurements. Saudi Med J. 2002 Nov;23(11):1367-72. PMID 12506298